CLINICAL TRIAL: NCT03761173
Title: FlowTriever All-Comer Registry for Patient Safety and Hemodynamics (FLASH)
Brief Title: FlowTriever All-Comer Registry for Patient Safety and Hemodynamics
Acronym: FLASH
Status: Completed | Type: Observational
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-002
Record Dates: First submitted 2018-11-28; First posted 2018-12-03 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: PE - Pulmonary Embolism; PE - Pulmonary Thromboembolism
Keywords: PE; pulmonary embolism; thromboembolism; thrombectomy; FlowTriever; Anticoagulation Medication
MeSH Terms: conditions — Pulmonary Embolism; Thromboembolism | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FlowTriever: Mechanical thrombectomy for pulmonary embolism
  Interventions: Device: FlowTriever System
- Conservative Therapy Sub-Study: Anticoagulation medication for pulmonary embolism (as directed by treating physician)
  Interventions: Drug: Anticoagulation Agents

INTERVENTIONS:
Device: FlowTriever System — Thrombectomy
  Groups: FlowTriever
Drug: Anticoagulation Agents — Anticoagulation medication
  Groups: Conservative Therapy Sub-Study

SUMMARY:
To evaluate the safety and effectiveness of the FlowTriever System for use in the removal of emboli from the pulmonary arteries in the treatment of acute pulmonary embolism (PE). The use of the device will be assessed in a real-world population, with eligibility criteria that closely approximate its use in clinical practice.

Up to 300 additional patients with anticoagulation treatment as the initial planned primary treatment strategy for intermediate risk PE will also be evaluated (US only).

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms consistent with acute PE
* Echo, CTPA or pulmonary angiographic evidence of proximal filling defect in at least one main or lobar pulmonary artery
* Scheduled for PE treatment with the FlowTriever System per the Investigator's discretion*

  * US only: Patients enrolled in the Conservative Therapy Sub-study are not required to meet this inclusion criteria but must instead be scheduled for primary anticoagulation therapy as the primary treatment strategy.

Exclusion Criteria:

* Unable to be anticoagulated with heparin or alternative
* Diagnosis with a minor PE with a less than 0.9 RV/LV ratio
* Known sensitivity to radiographic contrast agents that, in the Investigator's opinion, cannot be adequately pre-treated*
* Imaging evidence or other evidence that suggests, in the Investigator's opinion, the subject is not appropriate for mechanical thrombectomy intervention*
* Life expectancy < 30 days, as determined by Investigator
* Current participation in another investigational drug or device treatment study that, in the Investigator's opinion, would interfere with participation in this study

  * US Only Patients enrolled in the Conservative Therapy Sub-study are not required to meet these exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring treatment for pulmonary embolism.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catalin Toma, MD, Principal Investigator — University of Pittsburgh
Locations (81):
- United States (59):
  - UAB Division of Cardiovascular Disease, Birmingham, Alabama
  - University of Arizona College of Medicine, Tucson, Arizona
  - Pima Heart and Vascular, Tucson, Arizona
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Lakeland Vascular Institute, Lakeland, Florida
  - Palmetto General Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - Mount Sinai Medical Center of Florida, Miami, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Emory University, Atlanta, Georgia
  - Rush Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Javon Bea Hospital, Rockford, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Norton Healthcare, Louisville, Kentucky
  - Baptist Health Lousville, Louisville, Kentucky
  - Opelousas General, Opelousas, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - Ascension Genesys Hospital, Grand Blanc, Michigan
  - Ascension Providence Hospital, Madison Heights, Michigan
  - Ascension Providence Rochester Hospital, Rochester, Michigan
  - Beaumont Health, Royal Oak, Michigan
  - St. Joseph Mercy, Ypsilanti, Michigan
  - Metropolitan Heart and Vascular Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - University of Missouri, Columbia, Columbia, Missouri
  - Saint Luke's Hospital of Kansas City, Lee's Summit, Missouri
  - Valley Health, Ridgewood, New Jersey
  - Albany Medical Center, Albany, New York
  - SUNY, The University at Buffalo, Buffalo, New York
  - Northwell Health, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai, New York, New York
  - Jamaica Hospital, Queens, New York
  - St. Francis Hospital & Heart Center, Roslyn, New York
  - Westchester Medical Center, Valhalla, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Lexington Medical Center, West Columbia, South Carolina
  - Methodist Healthcare Foundation, Germantown, Tennessee
  - UTMC Knoxville, Knoxville, Tennessee
  - St. Thomas West, Nashville, Tennessee
  - CardioVoyage, Denison, Texas
  - Inova Fairfax, Falls Church, Virginia
  - Sentara, Norfolk, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Providence Sacred Heart, Spokane, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Allgemeines Krankenhaus AKH Wien, Vienna, Austria
- Belgium (2):
  - UZ Antwerpen, Antwerp
  - UZ Brussel, Brussels
- France (6):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Hopital de la Cavale Blanche - CHU Brest, Brest
  - CHU Grenoble, Grenoble
  - Institut Coeur Poumon - CHU de Lille, Lille
  - HCL Hôpital Louis Pradel - Hôpital Cardiologique, Lyon
  - European Hospital Georges Pompidou, Paris
- Germany (5):
  - Charité Hospital - Campus Virchow-Klinikum, Berlin
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - University Hospital, Heidelberg
  - Universitatsklinikum des Saarlandes, Homburg
  - Helios Kliniken Schwerin, Schwerin
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Spain (2):
  - Hospital Clínico San Carlos, Madrid
  - Gregorio Maranon University Hospital, Madrid
- Switzerland (3):
  - Inselspital, Bern
  - Kantonsspital Sankt Gallen, Sankt Gallen
  - Unispital, Zurich
- United Kingdom (2):
  - The Royal Free Hospital, London
  - The Royal London Hospital, Bart's Health, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Horowitz JM, Jaber WA, Stegman B, Rosenberg M, Fanola C, Bhat AP, Gondi S, Castle J, Ahmed M, Brown MA, Amin R, Bisharat M, Butros P, DuCoffe A, Savin M, Pollak JS, Weinberg MD, Brancheau D, Toma C. Mechanical Thrombectomy for High-Risk Pulmonary Embolism: Insights From the US Cohort of the FLASH Registry. J Soc Cardiovasc Angiogr Interv. 2023 Oct 31;3(1):101124. doi: 10.1016/j.jscai.2023.101124. eCollection 2024 Jan. PMID 39131977
- [Background] Khandhar S, Jaber W, Bunte MC, Cho K, Weinberg MD, Mina B, Stegman B, Pollak J, Khosla A, Elmasri F, Zlotnick D, Brancheau D, Koenig G, Bisharat M, Li J, Toma C. Longer-Term Outcomes Following Mechanical Thrombectomy for Intermediate- and High-Risk Pulmonary Embolism: 6-Month FLASH Registry Results. J Soc Cardiovasc Angiogr Interv. 2023 May 19;2(4):101000. doi: 10.1016/j.jscai.2023.101000. eCollection 2023 Jul-Aug. PMID 39131661
- [Background] Bangalore S, Horowitz JM, Beam D, Jaber WA, Khandhar S, Toma C, Weinberg MD, Mina B. Prevalence and Predictors of Cardiogenic Shock in Intermediate-Risk Pulmonary Embolism: Insights From the FLASH Registry. JACC Cardiovasc Interv. 2023 Apr 24;16(8):958-972. doi: 10.1016/j.jcin.2023.02.004. PMID 37100559
- [Background] Toma C, Jaber WA, Weinberg MD, Bunte MC, Khandhar S, Stegman B, Gondi S, Chambers J, Amin R, Leung DA, Kado H, Brown MA, Sarosi MG, Bhat AP, Castle J, Savin M, Siskin G, Rosenberg M, Fanola C, Horowitz JM, Pollak JS. Acute outcomes for the full US cohort of the FLASH mechanical thrombectomy registry in pulmonary embolism. EuroIntervention. 2023 Feb 20;18(14):1201-1212. doi: 10.4244/EIJ-D-22-00732. PMID 36349702
- [Background] Toma C, Bunte MC, Cho KH, Jaber WA, Chambers J, Stegman B, Gondi S, Leung DA, Savin M, Khandhar S, Kado H, Koenig G, Weinberg M, Beasley RE, Roberts J, Angel W, Sarosi MG, Qaqi O, Veerina K, Brown MA, Pollak JS. Percutaneous mechanical thrombectomy in a real-world pulmonary embolism population: Interim results of the FLASH registry. Catheter Cardiovasc Interv. 2022 Mar;99(4):1345-1355. doi: 10.1002/ccd.30091. Epub 2022 Feb 3. PMID 35114059

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FlowTriever
Started | 1000
Completed | 758
Not Completed | 242
Not completed — Lost to Follow-up | 93
Not completed — Withdrawal by Subject | 74
Not completed — Death | 45
Not completed — Withdrawal for Other Reasons | 29
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | FlowTriever
Number analyzed (Participants) | 999
Age, Categorical [Count of Participants; unit: Participants] — Population: Data was missing for one subject.
  Participants
    number analyzed (Participants) | 998
    <=18 years | 0
    Between 18 and 65 years | 547
    >=65 years | 451
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data was missing for one subject.
  years
    number analyzed (Participants) | 998
    (all) | 61.6 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 453
  Male | 546
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 698
  Unknown or Not Reported | 281
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 192
  White | 572
  More than one race | 1
  Unknown or Not Reported | 227
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: Data was missing for four subjects.
  kg/m^2
    number analyzed (Participants) | 995
    (all) | 33.8 (8.1)
Prior History of PE [Count of Participants; unit: Participants]
  Yes | 101
  No | 898
PE Classification [Count of Participants; unit: Participants] — Classifications are defined in 2019 European Society of Cardiology Guidelines for the Diagnosis and Management of Acute Pulmonary Embolism. Population: Data was missing for two subjects.
  Participants
    number analyzed (Participants) | 997
    High Risk | 143
    Intermediate-High Risk | 718
    Intermediate-Low Risk | 65
    Intermediate Risk, Not Further Classified | 71
Prior History of DVT [Count of Participants; unit: Participants] — Population: Data was missing for one subject.
  Participants
    number analyzed (Participants) | 998
    Yes | 187
    No | 811
Concomitant DVT [Count of Participants; unit: Participants] — Population: Data was missing for 10 subjects.
  Participants
    number analyzed (Participants) | 989
    Yes | 621
    No | 368
DVT Location [Count of Participants; unit: Participants] — Population: Data was collected for subjects with Concomitant DVT. Data was missing for eight subjects.
  Participants
    number analyzed (Participants) | 613
    Proximal Only | 209
    Distal Only | 308
    Both | 96
History of Cancer [Count of Participants; unit: Participants]
  Yes | 210
  No | 789
Active Cancer [Count of Participants; unit: Participants] — Population: Active cancer was collected for subjects with cancer history.
  Participants
    number analyzed (Participants) | 210
    Yes | 94
    No | 116
Lytic Contraindication [Count of Participants; unit: Participants] — Population: Data was missing for one subject.
  Participants
    number analyzed (Participants) | 998
    Yes | 303
    No | 695

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Major Adverse Events
Description: MAEs are defined as a composite, when one or more of the following events occur:
  * Device-related mortality through 48 hours after the index procedure, or
  * Major bleeding through 48 hours after the index procedure, or
  * Intra-procedural device-related or procedure-related adverse events, including:
    * Clinical deterioration defined by hemodynamic or respiratory worsening, or
    * Device-related pulmonary vascular injury, or
    * Device-related cardiac injury
  The components of the composite MAE endpoint were adjudicated by the independent Medical Monitor.
Time Frame: 48-hours after index procedure
Population: Full Analysis Population - all subjects who enrolled in the FLASH Study and met the inclusion and exclusion criteria. Outcome was not evaluable for 11 subjects, yielding 988 analyzed subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever
Number analyzed (Participants) | 988
Participants
  Yes | 24
  No | 964

2. Secondary Outcome: Device-Related Mortality
Description: Rate of subjects with device related mortality through 48 hours post index procedure
Time Frame: 48-hours after the index procedure
Population: Full Analysis Population - all subjects who enrolled in the FLASH Study and met the inclusion and exclusion criteria. Outcome was not evaluable for 13 subjects, yielding 986 analyzed subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever
Number analyzed (Participants) | 986
Participants
  Yes | 0
  No | 986

3. Secondary Outcome: Major Bleeding
Description: Rate of subjects with major bleeding through 48 hours after the index procedure (fatal bleeding; symptomatic bleeding in a critical area or organ; bleeding causing a fall in hemoglobin of ≥5 g/dL or leading to transfusion of 2 or more units of blood products)
Time Frame: 48 hours after index procedure
Population: Full Analysis Population - all subjects who enrolled in the FLASH Study and met the inclusion and exclusion criteria. Outcome was not evaluable for 12 subjects, yielding 987 analyzed subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever
Number analyzed (Participants) | 987
Participants
  Yes | 17
  No | 970

4. Secondary Outcome: Intraprocedural Device-related or Procedure-related Adverse Events
Description: Intraprocedural Device-related or procedure-related adverse events, including:
  * Clinical deterioration defined by hemodynamic or respiratory worsening, or
  * Device-related pulmonary vascular injury, or
  * Device-related cardiac injury.
Time Frame: Intraprocedural - occurring during the procedure or within 30 minutes of the FlowTriever Catheter being removed from the patient.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | FlowTriever
Number analyzed (Participants) | 987
Participants
  Yes | 8
  No | 979

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment through 6 months visit or study exit, if exited early.
Description: Reportable AEs include all events considered in the safety analyses (e.g., major bleedings), all device- and/or procedure-related AEs, as well as any event resulting in mortality. Events were adjudicated by independent medical monitor.
  Note: 196 patients had unknown mortality status due to early withdrawal or loss to follow-up before completing study visits as planned. The all-cause mortality rate at study exit among patients with confirmed mortality status was 5.6% (45/803).
Arm/Group | FlowTriever
All-Cause Mortality (participants affected / at risk) | 45/999
Serious Adverse Events (participants affected / at risk) | 125/999
Other Adverse Events (participants affected / at risk) | 0/999
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FlowTriever (N=999)
Pulmonary Embolism (Vascular disorders) | 12
Deep Vein Thrombosis (Vascular disorders) | 6
Haemodynamic Instability (Vascular disorders) | 3
Haemorrhage (Vascular disorders) | 3
Ischaemic Stroke (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2
Retroperitoneal Haematoma (Vascular disorders) | 2
Shock Haemorrhagic (Vascular disorders) | 2
Atrial Thombosis (Vascular disorders) | 1
Coronary Artery Stenosis (Vascular disorders) | 1
Hypovolaemic Shock (Vascular disorders) | 1
Intra-Abdominal Haematoma (Vascular disorders) | 1
Leriche Syndrome (Vascular disorders) | 1
Peripheral Ischaemia (Vascular disorders) | 1
Post Procedural Pulmonary Embolism (Vascular disorders) | 1
Retroperitoneal Haemorrhage (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Subarachnoid Haemorrhage (Vascular disorders) | 1
Syncope (Vascular disorders) | 1
Vasoplegia Syndrome (Vascular disorders) | 1
Cardiac Arrest (Cardiac disorders) | 5
Bradycardia (Cardiac disorders) | 3
Cardio-Respiratory Arrest (Cardiac disorders) | 3
Cardiac Failure (Cardiac disorders) | 2
Acute Pulmonary Oedema (Cardiac disorders) | 1
Aortic Valve Stenosis (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Bundle Branch Block, Left (Cardiac disorders) | 1
Cardiac Failure, Congestive (Cardiac disorders) | 1
Chest Discomfort (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 5
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 3
Subdural Haematoma (Injury, poisoning and procedural complications) | 2
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 2
Cardiac Procedure Complication (Injury, poisoning and procedural complications) | 1
Cardiac Valve Rupture (Injury, poisoning and procedural complications) | 1
Contrast Media Toxicity (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Vascular Access Site Complication (Injury, poisoning and procedural complications) | 1
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colorectal Cancer Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mallignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic Carcinoma, Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Cancer, Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Influenza (Respiratory, thoracic and mediastinal disorders) | 1
Lower Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia Pneumococcal (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal Injury (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 8
Blood Loss Anaemia (Blood and lymphatic system disorders) | 2
Heparin-induced Thrombocytopenia (Blood and lymphatic system disorders) | 2
Plasma Cell Myeloma (Blood and lymphatic system disorders) | 2
Death (General disorders) | 3
Multiple Organ Dysfunction Syndrome (General disorders) | 3
Septic Shock (Infections and infestations) | 2
Groin Abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Colon Cancer (Gastrointestinal disorders) | 1
Intestinal Perforation (Gastrointestinal disorders) | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1
Metabolic Encephalopathy (Nervous system disorders) | 1
Haemoglobin Decreased (Investigations) | 1
Mental Status Change (Psychiatric disorders) | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1
Arterial Repair (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03761173/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT03761173/SAP_001.pdf